CLINICAL TRIAL: NCT05681936
Title: Functional and Structural Changes in the Central Nervous System Following Spinal Cord Injury
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2022-00558
Record Dates: First submitted 2022-10-31; First posted 2023-01-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder Dysfunction; Degenerative Cervical Spinal Stenosis
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cross-sectional study: healthy controls
- Cross-sectional study: chronic traumatic SCI patients
- Cross-sectional study: non-traumatic SCI patients with degenerative spondylotic myelopathy
- Longitudinal study: healthy controls
- Longitudinal study: acute traumatic SCI patients (< 2 months after SCI)
- Longitudinal study: patients with neurogenic lower urinary tract dysfunction

SUMMARY:
Building on recent improvements, state-of-the-art functional MRI will be applied as an advanced diagnostic tool for the lumbosacral cord in spinal cord injury (SCI) patients to characterize the remaining neuronal activity of the motor and sensory neurons. Alterations in the activity pattern will reveal the effect upon task-related spinal cord activity of the lower motor neurons and sensory neurons undergoing trauma-induced neurodegeneration, at a spatial specificity that has not been possible so far. Results of this study will be of crucial importance because SCI patients can only profit from regeneration-inducing therapies if spinal neuronal function is preserved below the level of lesion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Informed consent
* Willing to take part and follow requirements of the protocol

Patients additionally need to fulfil the following study-specific inclusion criteria:

Cross-sectional study:

* Chronic traumatic SCI (> 12 months after injury) or
* Diagnosed degenerative spondylotic myelopathy (DCM)

Longitudinal study:

* Acute traumatic SCI (< 2 months after injury) or
* Patients with neurogenic lower urinary tract dysfunction (NLUTD) who undergo routine tibial nerve stimulation (TNS) treatment as part of their rehabilitation (but independently of this study) at Balgrist University Hospital

Exclusion Criteria:

* Age < 18 years
* Contraindications for MRI (presence of pacemaker or other type of stimulator in the body, presence of metallic foreign body in or on the body, etc.); we will comply with the imaging center's (SCMI) guidelines and in case of doubt we will exclude the participant from the study
* No informed consent
* History of psychiatric or neurological disease, apart from those induced by SCI (e.g.epilepsy)
* History of skull opening or head trauma
* Known or suspected non-adherence, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Women who are pregnant (when uncertain, participants will undergo urine testing) or breastfeeding
* Intention to become pregnant during the course of the study
* Body mass index (BMI) > 35
* Individuals especially in need of protection (according to Research with Human Subjects published by the Swiss Academy of Medical Sciences)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from the primary care clinic as well as via flyers distributed at hospital waiting rooms and patient support organisations.
  Healthy controls will be recruited via public announcements and via flyers distributed at the primary care clinic and two universities.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional study: lumbosacral functional fMRI | Baseline only
  Activations in the gray matter of the lumbosacral cord, as a response to sensory, motor, and somatosensory stimulations, or no stimulation (resting state). Spatiotemporal components of the BOLD signal as well as the couplings and anti-couplings between these components
Longitudinal study: lumbosacral functional fMRI | Change from baseline at 2-month, 6-month, and 12-month
  Activations in the gray matter of the lumbosacral cord, as a response to sensory, motor, and somatosensory stimulations, or no stimulation (resting state). Spatiotemporal components of the BOLD signal as well as the couplings and anti-couplings between these component
Cross-sectional study: brain functional MRI | Baseline only
  Activations in the cortical and subcortical areas of the brain as a response to sensory, motor, and somatosensory stimulations, or no stimulation (resting state)
Longitudinal study: brain functional MRI | Change from baseline at 2-month, 6-month, and 12-month
  Activations in the cortical and subcortical areas of the brain as a response to sensory, motor, and somatosensory stimulations, or no stimulation (resting state)

SECONDARY OUTCOMES:
Cross-sectional study: diffusion MRI in the spinal cord | Baseline only
  Directional diffusivities in the spinal cord (units of mm2/s)
Cross-sectional study: diffusion MRI in the spinal cord | Baseline only
  Fractional anisotropy in the spinal cord (unitless)
Longitudinal study: diffusion MRI in the spinal cord | Change from baseline at 2-month, 6-month, and 12-month
  Directional diffusivities in the spinal cord, measured (units of mm2/s)
Longitudinal study: diffusion MRI in the spinal cord | Change from baseline at 2-month, 6-month, and 12-month
  Fractional anisotropy in the spinal cord (unitless)
Cross-sectional study: structural MRI in spinal cord | Baseline only
  Cross-sectional areas of the spinal cord gray and white matter (units of mm2)
Longitudinal study: structural MRI in spinal cord | Change from baseline at 2-month, 6-month, and 12-month
  Cross-sectional areas of the spinal cord gray and white matter (units of mm2)
Cross-sectional study: magnetic resonance neurography of the lumbosacral plexus | Baseline only
  Thickness of nerves and nerve roots (units of mm2)
Cross-sectional study: magnetic resonance neurography of the lumbosacral plexus | Baseline only
  Nerve entry points into the spinal cord (for determining neurological levels)
Longitudinal study: magnetic resonance neurography of the lumbosacral plexus | Change from baseline at 2-month, 6-month, and 12-month
  Thickness of nerves and nerve roots (units of mm2)
Longitudinal study: magnetic resonance neurography of the lumbosacral plexus | Change from baseline at 2-month, 6-month, and 12-month
  Nerve entry points into the spinal cord (for determining neurological levels)
Cross-sectional study: diffusion MRI in the brain | Baseline only
  Directional diffusivities in the brain (units of mm2/s)
Cross-sectional study: diffusion MRI in the brain | Baseline only
  Fractional anisotropy in the brain (unitless)
Longitudinal study: diffusion MRI in the brain | Change from baseline at 2-month, 6-month, and 12-month
  Directional diffusivities in the brain (units of mm2/s)
Longitudinal study: diffusion MRI in the brain | Change from baseline at 2-month, 6-month, and 12-month
  Fractional anisotropy in the brain (unitless)
Cross-sectional study: structural MRI in the brain | Baseline only
  Cortical thickness (units of mm)
Cross-sectional study: structural MRI in the brain | Baseline only
  Volumes of the brain gray and white matter (units of mm3)
Longitudinal study: structural MRI in the brain | Change from baseline at 2-month, 6-month, and 12-month
  Cortical thickness (units of mm)
Longitudinal study: structural MRI in the brain | Change from baseline at 2-month, 6-month, and 12-month
  Volumes of the brain gray and white matter (units of mm3)
Cross-sectional study: nerve conduction study | Baseline only
  Latencies of F waves (units of ms). Period between initial stimulation and F wave elicitation in the tibial and peroneal motor nerves.
Cross-sectional study: nerve conduction study | Baseline only
  Amplitudes of F waves in the tibial and peroneal motor nerves (units of microV)
Cross-sectional study: nerve conduction study | Baseline only
  Duration of F waves in the tibial and peroneal motor (units of ms)
Longitudinal study: nerve conduction study | Change from baseline at 2-month, 6-month, and 12-month
  Latencies of F waves (units of ms). Period between initial stimulation and F wave elicitation in the tibial and peroneal motor nerves.
Longitudinal study: nerve conduction study | Change from baseline at 2-month, 6-month, and 12-month
  Amplitudes of F waves in the tibial and peroneal motor nerves (units of microV)
Longitudinal study: nerve conduction study | Change from baseline at 2-month, 6-month, and 12-month
  Duration of F waves in the tibial and peroneal motor (units of ms)
Cross-sectional study: motor evoked potentials (MEP) | Baseline only
  Latencies (units of ms)
Cross-sectional study: motor evoked potentials (MEP) | Baseline only
  Amplitudes (units of mV)
Longitudinal study: motor evoked potentials (MEP) | Change from baseline at 2-month, 6-month, and 12-month
  Latencies (units of ms)
Longitudinal study: motor evoked potentials (MEP) | Change from baseline at 2-month, 6-month, and 12-month
  Amplitudes (units of mV)
Cross-sectional study: American Spinal Injury Association Impairment Scale (AIS) from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Baseline only
  AIS quantifies the severity of the spinal cord injury. AIS (ASIA Impairment Scale) grades from A-E, whereas grade A (complete spinal cord injury) is worse than grade E (no impairment)
Cross-sectional study: Lower Extremities Motor Scale (LEMS) from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Baseline only
  LEMS is based on assessments of ISNCSCI and composed from the sum of muscle function grading of the five key muscles of the lower limbs. It consists of a 6-point scale (0=no; 5=normal activity) for each muscle and body site. The lowest possible score in the total LEMS score for one body site is 0 (symptomatic); the highest possible score is 50 (asymptomatic)
Cross-sectional study: Upper Extremities Motor Scale (UEMS) from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Baseline only
  UEMS is based on assessments of ISNCSCI and composed from the sum of muscle function grading of the five key muscles of the upper limbs. It consists of a 6-point scale (0=no; 5=normal activity) for each muscle and body site. The lowest possible score in the total UEMS score for one body site is 0 (symptomatic); the highest possible score is 50 (asymptomatic)
Cross-sectional study: Light touch (LT) score from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Baseline only
  The LT score is based on assessments of ISNCSCI and represents the sum of sensory function of 28 dermatome pairs in terms of light touch sensation. It consists of a 2-point scale (0=absent sensation; 1=altered (impaired or partial sensation, including hyperesthesia); 2 = normal or intact sensation) for each dermatome and body site. The lowest and highest possible LT score for one body site is 0 and 56, respectively
Cross-sectional study: Pin prick (PP) score from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Baseline only
  The PP score is based on assessments of ISNCSCI and represents the sum of sensory function of 28 dermatome pairs in terms of pin prick discrimination. It consists of a 2-point scale (0=absent discrimination; 1=altered (impaired or partial discrimination); 2 = normal or intact discrimination) for each dermatome and body site. The lowest and highest possible PP score for one body site is 0 and 56, respectively
Longitudinal study: American Spinal Injury Association Impairment Scale (AIS) from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Change from baseline at 2-month, 6-month, and 12-month
  AIS quantifies the severity of the spinal cord injury. AIS (ASIA Impairment Scale) grades from A-E, whereas grade A (complete spinal cord injury) is worse than grade E (no impairment).
Longitudinal study: Lower Extremities Motor Scale (LEMS) from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Change from baseline at 2-month, 6-month, and 12-month
  LEMS is based on assessments of ISNCSCI and composed from the sum of muscle function grading of the five key muscles of the lower limbs. It consists of a 6-point scale (0=no; 5=normal activity) for each muscle and body site. The lowest possible score in the total LEMS score for one body site is 0 (symptomatic); the highest possible score is 50 (asymptomatic)
Longitudinal study: Upper Extremities Motor Scale (UEMS) from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Change from baseline at 2-month, 6-month, and 12-month
  UEMS is based on assessments of ISNCSCI and composed from the sum of muscle function grading of the five key muscles of the upper limbs. It consists of a 6-point scale (0=no; 5=normal activity) for each muscle and body site. The lowest possible score in the total UEMS score for one body site is 0 (symptomatic); the highest possible score is 50 (asymptomatic)
Longitudinal study: Light touch (LT) score from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Change from baseline at 2-month, 6-month, and 12-month
  The LT score is based on assessments of ISNCSCI and represents the sum of sensory function of 28 dermatome pairs in terms of light touch sensation. It consists of a 2-point scale (0=absent sensation; 1=altered (impaired or partial sensation, including hyperesthesia); 2 = normal or intact sensation) for each dermatome and body site. The lowest and highest possible LT score for one body site is 0 and 56, respectively
Longitudinal study: Pin prick (PP) score from the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Change from baseline at 2-month, 6-month, and 12-month
  The PP score is based on assessments of ISNCSCI and represents the sum of sensory function of 28 dermatome pairs in terms of pin prick discrimination. It consists of a 2-point scale (0=absent discrimination; 1=altered (impaired or partial discrimination); 2 = normal or intact discrimination) for each dermatome and body site. The lowest and highest possible PP score for one body site is 0 and 56, respectively
Cross-sectional study: Graded and Redefined Assessment of Strength, Sensation and Prehension (GRASSP) | Baseline only
  GRASSP measures sensorimotor and prehension function through three domains (strength, sensation and prehension) which are important in describing arm and hand function. The total GRASSP score ranges from 0 to 116 points, where a higher score indicates a better outcome
Longitudinal study: Graded and Redefined Assessment of Strength, Sensation and Prehension (GRASSP) | Change from baseline at 2-month, 6-month, and 12-month
  GRASSP measures sensorimotor and prehension function through three domains (strength, sensation and prehension) which are important in describing arm and hand function. The total GRASSP score ranges from 0 to 116 points, where a higher score indicates a better outcome
Cross-sectional study: European Multicenter Study about SCI (EMSCI) pain questionnaire | Baseline only
  The EMSCI pain questionnaire rates various aspects of pain (e.g., current pain intensity, mean and maximal pain intensity during the last week before the assessment, location and quality of pain, intensity of allodynia and paresthesia). Pain intensity is quantified on an 11-point numeric scale (0=no pain; 10=worst imaginable pain)
Longitudinal study: European Multicenter Study about SCI (EMSCI) pain questionnaire | Change from baseline at 2-month, 6-month, and 12-month
  The EMSCI pain questionnaire rates various aspects of pain (e.g., current pain intensity, mean and maximal pain intensity during the last week before the assessment, location and quality of pain, intensity of allodynia and paresthesia). Pain intensity is quantified on an 11-point numeric scale (0=no pain; 10=worst imaginable pain)
Cross-sectional study: sympathetic skin response including hand, sole and perineum recordings | Baseline only
  Latencies (units of ms)
Cross-sectional study: sympathetic skin response including hand, sole and perineum recordings | Baseline only
  Amplitudes (units of microV)
Longitudinal study: sympathetic skin response including hand, sole and perineum recordings | Change from baseline at 2-month, 6-month, and 12-month
  Latencies (units of ms)
Longitudinal study: sympathetic skin response including hand, sole and perineum recordings | Change from baseline at 2-month, 6-month, and 12-month
  Amplitudes (units of microV)
Cross-sectional study: Spinal Cord Independence Measure (SCIM III) | Baseline only
  The SCIM-III ("Spinal Cord Independence Measure III") score is based on questions concerning independence of persons with a spinal cord injured. It consists of 19 items covering 3 domains, self-care, respiration and sphincter management, and mobility. The self-care subscale ranges from 0 to 20. The respiration and sphincter management subscale ranges from 0 to 40. The mobility subscale ranges from 0 to 40. Total score ranges from 0 (symptomatic) to 100 (asymptomatic). Higher scores reflect higher levels of independence.
Longitudinal study: Spinal Cord Independence Measure (SCIM III) | Change from baseline at 2-month, 6-month, and 12-month
  The SCIM-III ("Spinal Cord Independence Measure III") score is based on questions concerning independence of persons with a spinal cord injured. It consists of 19 items covering 3 domains, self-care, respiration and sphincter management, and mobility. The self-care subscale ranges from 0 to 20. The respiration and sphincter management subscale ranges from 0 to 40. The mobility subscale ranges from 0 to 40. Total score ranges from 0 (symptomatic) to 100 (asymptomatic). Higher scores reflect higher levels of independence
Cross-sectional study: Walking index for Spinal Cord Injury (WISCI) | Baseline only
  WISCI is an ordinal 20-point scale (0=unable to stand and/or participate in walking; 20=ambulates with no devices, with brace and no assistance) to assess walking function
Longitudinal study: Walking index for Spinal Cord Injury (WISCI) | Change from baseline at 2-month, 6-month, and 12-month
  WISCI is an ordinal 20-point scale (0=unable to stand and/or participate in walking; 20=ambulates with no devices, with brace and no assistance) to assess walking function
Longitudinal study: International Prostate Symptom Score (IPSS) (only in patients with neurogenic lower urinary tract dysfunction) | Change between baseline and follow-up (6-12 weeks of tibial nerve stimulation)
  The IPSS score is based on questions concerning urinary symptoms and quality of life (QoL). It consists of 8 items covering 7 urinary symptoms related dimensions (subscales) and 1 additional item assessing quality of life. Each item is rated on a 6-point scale (0=not at all; 5=almost always). The lowest possible score in the total IPSS score is 0 (asymptomatic); the highest possible score is 35 (symptomatic). The QoL index is rated on a 7-point scale, with 0 indicating "delighted" and 6 "terrible"
Longitudinal study: Qualiveen questionnaire (only in patients with neurogenic lower urinary tract dysfunction) | Change between baseline and follow-up (6-12 weeks of tibial nerve stimulation)
  Qualiveen-30 assesses the Specific Impact of Urinary Problems (SIUP) on Quality of Life. It consists of 30 items covering 4 domains, namely inconvenience (9 questions), restrictions (8 questions), fears (8 questions), and impact on daily life (5 questions). Each item is rated on a 5-point ordinal scale (0=asymptomatic; 4=symptomatic). The index of the SIUP on Quality of Life is the mean of the four individual scores. The lowest possible overall score in the Qualiveen-30 is 0 (Urinary problems have no specific impact on QoL); the highest possible score is 30 (Urinary problems have a huge specific impact on QoL)
Longitudinal study: Urinary Symptom Profile (USP) (only in patients with neurogenic lower urinary tract dysfunction) | Change between baseline and follow-up (6-12 weeks of tibial nerve stimulation)
  The USP score is based on questions concerning urinary symptoms and their severity in males and females. It consists of 13 items covering 3 dimensions (subscales) with 7 overactive bladder (OAB), 3 stress urinary incontinence (SUI), and 3 low stream (LS) related items. Each item is rated on a 4-point scale. The lowest score is 0 (asymptomatic); the highest score is 3 (symptomatic)
Longitudinal study: Overactive Bladder (ICIQ-OAB) questionnaire (only in patients with neurogenic lower urinary tract dysfunction) | Change between baseline and follow-up (6-12 weeks of tibial nerve stimulation)
  International Consultation on Incontinence Questionnaire Overactive Bladder Quality of Life ICIQ-OAB-QoL is a 26-item questionnaire evaluating quality of life (QoL) in patients with overactive bladder. Scores range from 25-160, with greater values indicating increased impact on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Freund, Prof. Dr. med. Dr. rer. nat., Principal Investigator — University of Zurich
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland